CLINICAL TRIAL: NCT00678210
Title: A Phase 2B, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Trial Evaluating The Efficacy And Safety Of Dose Regimens With Oral CP-690,550 In The Treatment Of Subjects With Moderate To Severe Chronic Plaque Psoriasis
Brief Title: Effectiveness and Safety of 3 Dosing Regimens of CP-690,550 to Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921047
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-11

CONDITIONS: Psoriasis
Keywords: dose response; PASI 75 response endpoint; subjects with moderate to severe chronic plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: CP-690,550
- 2 (Experimental)
  Interventions: Drug: CP-690,550
- 3 (Experimental)
  Interventions: Drug: CP-690,550
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-690,550 — tablets, 2 mg BID for 12 weeks
  Arms: 1
Drug: CP-690,550 — tablets, 5 mg BID for 12 weeks
  Arms: 2
Drug: CP-690,550 — tablets, 15 mg BID for 12 weeks
  Arms: 3
Drug: Placebo — tablets, BID for 12 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to determine the effectiveness and safety, over 12 weeks, of 3 dosing regimens of CP-690,550 for the treatment of adults with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with plaque psoriasis for at least 6 months.
* Have plaque psoriasis covering at least 15% of their total body.
* Be a candidate for phototherapy or systemic treatment of psoriasis (either naïve or history of previous treatment).
* Be willing and able to comply with scheduled visits, treatment plan and other study procedures.

Exclusion Criteria:

* Currently have non-plaque forms of psoriasis or drug-induced psoriasis.
* Subject cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot discontinue phototherapy.
* Subject is participating in another trial using an investigational agent or procedure.
* Women who are pregnant or breast-feeding or considering becoming pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (26):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, West Dundee, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, East Windsor, New Jersey
  - Pfizer Investigational Site, Paramus, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Lake Oswego, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Webster, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Norfolk, Virginia
- Canada (12):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, North Bay, Ontario
  - Pfizer Investigational Site, Waterloo, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec

REFERENCES:
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Valenzuela F, Papp KA, Pariser D, Tyring SK, Wolk R, Buonanno M, Wang J, Tan H, Valdez H. Effects of tofacitinib on lymphocyte sub-populations, CMV and EBV viral load in patients with plaque psoriasis. BMC Dermatol. 2015 May 8;15:8. doi: 10.1186/s12895-015-0025-y. PMID 25951857
- [Derived] Menter A, Papp KA, Tan H, Tyring S, Wolk R, Buonanno M. Efficacy of tofacitinib, an oral janus kinase inhibitor, on clinical signs of moderate-to-severe plaque psoriasis in different body regions. J Drugs Dermatol. 2014 Mar;13(3):252-6. PMID 24595567
- [Derived] Bushmakin AG, Mamolo C, Cappelleri JC, Stewart M. The relationship between pruritus and the clinical signs of psoriasis in patients receiving tofacitinib. J Dermatolog Treat. 2015 Feb;26(1):19-22. doi: 10.3109/09546634.2013.861891. Epub 2013 Dec 2. PMID 24289224
- [Derived] Strober B, Buonanno M, Clark JD, Kawabata T, Tan H, Wolk R, Valdez H, Langley RG, Harness J, Menter A, Papp K. Effect of tofacitinib, a Janus kinase inhibitor, on haematological parameters during 12 weeks of psoriasis treatment. Br J Dermatol. 2013 Nov;169(5):992-9. doi: 10.1111/bjd.12517. PMID 23855761
- [Derived] Papp KA, Menter A, Strober B, Langley RG, Buonanno M, Wolk R, Gupta P, Krishnaswami S, Tan H, Harness JA. Efficacy and safety of tofacitinib, an oral Janus kinase inhibitor, in the treatment of psoriasis: a Phase 2b randomized placebo-controlled dose-ranging study. Br J Dermatol. 2012 Sep;167(3):668-77. doi: 10.1111/j.1365-2133.2012.11168.x. PMID 22924949
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921047&StudyName=Effectiveness%20and%20safety%20of%203%20dosing%20regimens%20of%20CP-690%2C550%20to%20placebo%20in%20subjects%20with%20moderate%20to%20severe%20chronic%20plaque%20psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 2 mg: CP-690,550 tablets equivalent to CP-690,550 2 milligram (mg) orally twice daily for 12 weeks.
- CP-690,550 5 mg: CP-690,550 tablets equivalent to CP-690,550 5 mg orally twice daily for 12 weeks.
- CP-690,550 15 mg: CP-690,550 tablets equivalent to CP-690,550 15 mg orally twice daily for 12 weeks.
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily for 12 weeks.
Period: Overall Study
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Started | 49 | 49 | 49 | 50
Completed | 38 | 38 | 43 | 30
Not Completed | 11 | 11 | 6 | 20
Not completed — Adverse Event | 1 | 2 | 3 | 3
Not completed — Lack of Efficacy | 2 | 3 | 1 | 9
Not completed — Lost to Follow-up | 4 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4 | 1 | 7
Not completed — Other | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CP-690,550 2 mg: CP-690,550 tablets equivalent to CP-690,550 2 mg orally twice daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo | Total
Number analyzed (Participants) | 49 | 49 | 49 | 50 | 197
Age, Customized [Number; unit: participants]
  18 to 44 years | 23 | 25 | 28 | 20 | 96
  45 to 54 years | 13 | 14 | 10 | 18 | 55
  54 to 64 years | 9 | 9 | 6 | 10 | 34
  Greater than or equal to 65 years | 4 | 1 | 5 | 2 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 18 | 14 | 72
  Male | 29 | 29 | 31 | 36 | 125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a 75% Improvement in Psoriasis Area and Severity Index (PASI 75) Score at Week 12
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%) - 6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor(head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4).
Time Frame: Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of investigational drug and had at least 1 valid post-baseline efficacy assessment. Missing values were imputed using last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48 | 50
percentage of participants | 25.00 | 40.82 | 66.67 | 2.00

2. Secondary Outcome: Percentage of Participants Achieving Physician's Global Assessment (PGA) Score of "Clear" or "Almost Clear"
Description: Physician global assessment of psoriasis is global consideration of the erythema, induration and scaling across all psoriatic lesions, rated separately over the whole body according to a 5-point severity scale ranged from 0 to 4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. The severity scores are summed and averaged after which the total average is rounded to the nearest whole number score to determine the treatment area overall severity of psoriasis score and category. The score of 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe.
Time Frame: Week 2, 4, 8, 12, 14, 16
Population: FAS included all participants who received at least 1 dose of investigational drug and had at least 1 valid post-baseline efficacy assessment. Missing values imputed using LOCF for week 2, 4, 8, 12 and no imputation done for week 14, 16. n=participants evaluable for this measure at specified time points for each arm group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 50
percentage of participants
  Week 2 (n=48, 48, 48, 49) | 8.33 | 12.50 | 16.67 | 4.08
  Week 4 (n=49, 49, 48, 50) | 18.37 | 28.57 | 33.33 | 4.00
  Week 8 (n=49, 49, 48, 50) | 24.49 | 44.90 | 56.25 | 14.00
  Week 12 (n=49, 49, 48, 50) | 24.49 | 40.82 | 72.92 | 10.00
  Week 14 (n=38, 37, 37, 33) | 23.68 | 35.14 | 56.76 | 9.09
  Week 16 (n=37, 37, 41, 30) | 24.32 | 18.92 | 41.46 | 10.00

3. Secondary Outcome: Percentage of Participants Achieving a 75% Improvement in Psoriasis Area and Severity Index (PASI 75) Score
Description: as for outcome 1
Time Frame: Week 2, 4, 8, 14, 16
Population: FAS included all participants who received at least 1 dose of investigational drug and had at least 1 valid post-baseline efficacy assessment. Missing values imputed using LOCF for week 2, 4, 8 and no imputation done for week 14, 16. n=participants evaluable for this measure at specified time points for each arm group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48 | 50
percentage of participants
  Week 2 (n=47, 48, 48, 49) | 0.00 | 2.08 | 2.08 | 0.00
  Week 4 (n=48, 49, 48, 50) | 8.33 | 14.29 | 20.83 | 0.00
  Week 8 (n=48, 49, 48, 50) | 20.83 | 40.82 | 62.50 | 2.00
  Week 14 (n=38, 37, 37, 33) | 23.68 | 37.84 | 59.46 | 6.06
  Week 16 (n=37, 36, 41, 30) | 24.32 | 22.22 | 39.02 | 6.67

4. Secondary Outcome: Percentage of Participants Achieving a 50% Improvement in Psoriasis Area and Severity Index (PASI 50) Score
Description: as for outcome 1
Time Frame: Week 2, 4, 8, 12, 14, 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48 | 50
percentage of participants
  Week 2 (n=47, 48, 48, 49) | 10.64 | 14.58 | 25.00 | 0.00
  Week 4 (n=48, 49, 48, 50) | 29.17 | 44.90 | 62.50 | 6.00
  Week 8 (n=48, 49, 48, 50) | 41.67 | 55.10 | 79.17 | 14.00
  Week 12 (n=48, 49, 48, 50) | 39.58 | 65.31 | 87.50 | 20.00
  Week 14 (n=38, 37, 37, 33) | 42.11 | 59.46 | 86.49 | 24.24
  Week 16 (n=37, 36, 41, 30) | 40.54 | 47.22 | 68.29 | 23.33

5. Secondary Outcome: Percentage of Participants Achieving a 90% Improvement in Psoriasis Area and Severity Index (PASI 90) Score
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%)-6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4).
Time Frame: Week 12
Population: FAS included all participants who received at least 1 dose of investigational drug and had at least 1 valid post-baseline efficacy assessment. Missing values imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48 | 50
percentage of participants | 14.58 | 18.37 | 33.33 | 0.00

6. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Component Scores and Total Score
Description: as for outcome 5
Time Frame: Baseline, Week 2, 4, 8, 12, 14, 16
Population: FAS included all participants who received at least 1 dose of investigational drug and had at least 1 valid post-baseline efficacy assessment. No imputation was done. n=participants evaluable for this measure at specified time points for each arm group respectively.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48 | 50
units on a scale
  Baseline: Head/Neck Erythema (n=48, 49, 48, 50) | 2.1 (0.13) | 2.1 (0.14) | 2.4 (0.15) | 2.4 (0.12)
  Baseline: Upper Limbs Erythema (n=48, 49, 48, 50) | 2.8 (0.09) | 2.7 (0.11) | 2.8 (0.10) | 2.9 (0.07)
  Baseline: Trunk Erythema (n=48, 49, 48, 50) | 2.6 (0.13) | 2.6 (0.14) | 2.9 (0.10) | 2.8 (0.09)
  Baseline: Lower Limbs Erythema (n=48, 49, 48, 50) | 3.0 (0.08) | 2.9 (0.11) | 3.0 (0.11) | 3.1 (0.08)
  Week 2: Head/Neck Erythema (n=47, 48, 48, 49) | 1.8 (0.15) | 1.4 (0.14) | 1.4 (0.15) | 2.2 (0.12)
  Week 2: Upper Limbs Erythema (n=47, 48, 48, 49) | 2.2 (0.12) | 2.2 (0.13) | 2.0 (0.10) | 2.7 (0.09)
  Week 2: Trunk Erythema (n=47, 48, 48, 49) | 2.1 (0.14) | 2.0 (0.17) | 2.1 (0.14) | 2.7 (0.09)
  Week 2: Lower Limbs Erythema (n=47, 48, 48, 49) | 2.6 (0.11) | 2.4 (0.13) | 2.3 (0.14) | 2.9 (0.11)
  Week 4: Head/Neck Erythema (n=47, 47, 48, 46) | 1.5 (0.14) | 1.1 (0.15) | 1.0 (0.14) | 2.1 (0.15)
  Week 4: Upper Limbs Erythema (n=47, 47, 48, 46) | 1.9 (0.13) | 1.7 (0.14) | 1.5 (0.09) | 2.5 (0.11)
  Week 4: Trunk Erythema (n= 47, 47, 48, 46) | 1.8 (0.15) | 1.7 (0.17) | 1.6 (0.13) | 2.5 (0.11)
  Week 4: Lower Limbs Erythema (n= 47, 47, 48, 46) | 2.3 (0.13) | 2.0 (0.15) | 1.8 (0.13) | 2.8 (0.11)
  Week 8: Head/Neck Erythema (n=43, 40, 47, 39) | 1.2 (0.15) | 0.8 (0.16) | 0.6 (0.13) | 1.8 (0.18)
  Week 8: Upper Limbs Erythema (n=43, 40, 47, 39) | 1.6 (0.15) | 1.4 (0.14) | 1.1 (0.12) | 2.3 (0.12)
  Week 8: Trunk Erythema (n=43, 40, 47, 39) | 1.5 (0.16) | 1.3 (0.16) | 1.2 (0.16) | 2.3 (0.13)
  Week 8: Lower Limbs Erythema (n=43, 40, 47, 39) | 1.8 (0.14) | 1.4 (0.16) | 1.2 (0.14) | 2.5 (0.11)
  Week 12: Head/Neck Erythema (n=38, 39, 43, 34) | 1.1 (0.17) | 0.8 (0.15) | 0.4 (0.11) | 1.7 (0.19)
  Week 12: Upper Limbs Erythema (n=38, 39, 43, 34) | 1.5 (0.17) | 1.3 (0.12) | 1.0 (0.12) | 2.3 (0.15)
  Week 12: Trunk Erythema (n=38, 39, 43, 34) | 1.5 (0.18) | 1.1 (0.17) | 0.9 (0.16) | 2.4 (0.17)
  Week 12: Lower Limbs Erythema (n=38, 39, 43, 34) | 1.8 (0.17) | 1.3 (0.13) | 1.2 (0.15) | 2.6 (0.13)
  Week 14: Head/Neck Erythema (n=38, 37, 37, 33) | 1.2 (0.18) | 1.1 (0.14) | 0.9 (0.17) | 1.7 (0.20)
  Week 14: Upper Limbs Erythema (n=38, 37, 37, 33) | 1.8 (0.17) | 1.5 (0.16) | 1.3 (0.16) | 2.3 (0.14)
  Week 14: Trunk Erythema (n=38, 37, 37, 33) | 1.6 (0.19) | 1.4 (0.18) | 1.2 (0.20) | 2.4 (0.18)
  Week 14: Lower Limbs Erythema (n=38, 37, 37, 33) | 2.0 (0.17) | 1.6 (0.17) | 1.4 (0.18) | 2.6 (0.11)
  Week 16: Head/Neck Erythema (n=37, 36, 41, 30) | 1.3 (0.20) | 1.5 (0.16) | 1.0 (0.18) | 1.8 (0.22)
  Week 16: Upper Limbs Erythema (n=37, 36, 41, 30) | 1.9 (0.21) | 1.8 (0.14) | 1.7 (0.15) | 2.3 (0.14)
  Week 16: Trunk Erythema (n=37, 36, 41, 30) | 1.8 (0.21) | 1.8 (0.17) | 1.8 (0.18) | 2.3 (0.18)
  Week 16: Lower Limbs Erythema (n=37, 36, 41, 30) | 2.2 (0.18) | 1.8 (0.15) | 1.7 (0.18) | 2.7 (0.13)
  Baseline: Head/Neck Induration (n=48, 49, 48, 50) | 2.0 (0.14) | 1.8 (0.13) | 2.1 (0.15) | 2.0 (0.13)
  Baseline: Upper Limbs Induration(n=48, 49, 48, 50) | 2.5 (0.11) | 2.6 (0.11) | 2.7 (0.11) | 2.5 (0.10)
  Baseline: Trunk Induration (n=48, 49, 48, 50) | 2.4 (0.12) | 2.3 (0.12) | 2.6 (0.12) | 2.7 (0.09)
  Baseline: Lower Limbs Induration(n=48, 49, 48, 50) | 2.8 (0.09) | 2.7 (0.10) | 2.8 (0.12) | 2.7 (0.09)
  Week 2: Head/Neck Induration (n=47, 48, 48, 49) | 1.4 (0.15) | 1.4 (0.14) | 1.3 (0.15) | 1.9 (0.12)
  Week 2: Upper Limbs Induration(n=47, 48, 48, 49) | 2.0 (0.13) | 2.1 (0.12) | 1.9 (0.13) | 2.4 (0.10)
  Week 2: Trunk Induration (n=47, 47, 48, 46) | 2.1 (0.15) | 1.7 (0.15) | 2.0 (0.13) | 2.4 (0.11)
  Week 2: Lower Limbs Induration(n=47, 48, 48, 49) | 2.5 (0.12) | 2.4 (0.12) | 2.1 (0.14) | 2.6 (0.09)
  Week 4: Head/Neck Induration (n=47, 47, 48, 46) | 1.2 (0.14) | 0.8 (0.13) | 0.8 (0.14) | 1.7 (0.14)
  Week 4: Upper Limbs Induration (n=47, 47, 48, 46) | 1.9 (0.13) | 1.7 (0.13) | 1.4 (0.14) | 2.2 (0.12)
  Week 4: Trunk Induration (n=47, 47, 48, 46) | 1.7 (0.15) | 1.5 (0.15) | 1.4 (0.14) | 2.3 (0.11)
  Week 4: Lower Limbs Induration (n=47, 47, 48, 46) | 2.2 (0.14) | 1.9 (0.13) | 1.6 (0.14) | 2.3 (0.11)
  Week 8: Head/Neck Induration (n=43, 40, 47, 39) | 1.0 (0.14) | 0.6 (0.14) | 0.5 (0.13) | 1.5 (0.14)
  Week 8: Upper Limbs Induration (n=43, 40, 47, 39) | 1.7 (0.16) | 1.4 (0.14) | 1.2 (0.15) | 2.2 (0.12)
  Week 8: Trunk Induration (n=43, 40, 47, 39) | 1.5 (0.17) | 1.1 (0.17) | 1.1 (0.16) | 2.0 (0.13)
  Week 8: Lower Limbs Induration (n=43, 40, 47, 39) | 1.8 (0.17) | 1.3 (0.15) | 1.2 (0.16) | 2.2 (0.12)
  Week 12: Head/Neck Induration (n=38, 39, 43, 34) | 1.0 (0.17) | 0.5 (0.12) | 0.3 (0.10) | 1.5 (0.18)
  Week 12: Upper Limbs Induration (n=38, 37, 37, 33) | 1.4 (0.17) | 1.2 (0.12) | 1.0 (0.14) | 2.0 (0.16)
  Week 12: Trunk Induration (n=38, 39, 43, 34) | 1.4 (0.18) | 0.9 (0.16) | 0.8 (0.15) | 2.0 (0.17)
  Week 12: Lower limbs induration (n=38, 39, 43, 34) | 1.7 (0.17) | 1.2 (0.14) | 1.0 (0.14) | 2.2 (0.14)
  Week 14: Head/Neck Induration (n=38, 37, 37, 33) | 1.0 (0.16) | 0.9 (0.15) | 0.7 (0.16) | 1.4 (0.17)
  Week 14: Upper Limbs Induration (n=38, 37, 37, 33) | 1.8 (0.18) | 1.4 (0.16) | 1.3 (0.16) | 2.1 (0.14)
  Week 14: Trunk Induration (n=38, 37, 37, 33) | 1.4 (0.18) | 1.3 (0.18) | 1.1 (0.18) | 1.9 (0.17)
  Week 14: Lower Limbs Induration (n=38, 37, 37, 33) | 1.9 (0.16) | 1.5 (0.17) | 1.3 (0.18) | 2.2 (0.14)
  Week 16: Head/Neck Induration (n=37, 36, 41, 30) | 1.1 (0.18) | 1.2 (0.17) | 0.8 (0.15) | 1.6 (0.18)
  Week 16: Upper Limbs Induration (n=37, 36, 41, 30) | 1.8 (0.20) | 1.9 (0.16) | 1.5 (0.16) | 2.2 (0.15)
  Week 16: Trunk Induration (n=37, 36, 41, 30) | 1.5 (0.20) | 1.6 (0.18) | 1.5 (0.17) | 2.1 (0.18)
  Week 16: Lower Limbs Induration (n=37, 36, 41, 30) | 1.9 (0.19) | 1.8 (0.15) | 1.4 (0.17) | 2.4 (0.14)
  Baseline: Head/Neck Scaling (n=48, 49, 48, 50) | 2.1 (0.16) | 2.2 (0.13) | 2.3 (0.14) | 2.2 (0.14)
  Baseline: Upper Limbs Scaling (n=48, 49, 48, 50) | 2.5 (0.10) | 2.8 (0.11) | 2.6 (0.09) | 2.6 (0.10)
  Baseline: Trunk Scaling (n=48, 49, 48, 50) | 2.4 (0.14) | 2.4 (0.14) | 2.5 (0.12) | 2.6 (0.11)
  Baseline: Lower Limbs Scaling (n=48, 49, 48, 50) | 3.1 (0.10) | 2.9 (0.11) | 2.7 (0.12) | 2.9 (0.09)
  Week 2: Head/Neck Scaling (n=47, 48, 48, 49) | 1.7 (0.16) | 1.6 (0.16) | 1.4 (0.16) | 1.9 (0.13)
  Week 2: Upper Limbs Scaling (n=48, 49, 48, 50) | 2.1 (0.13) | 2.2 (0.13) | 2.0 (0.12) | 2.4 (0.11)
  Week 2: Trunk Scaling (n=47, 48, 48, 49) | 2.1 (0.14) | 1.8 (0.16) | 1.9 (0.12) | 2.3 (0.12)
  Week 2: Lower Limbs Scaling (n=47, 48, 48, 49) | 2.6 (0.12) | 2.5 (0.14) | 2.1 (0.13) | 2.7 (0.11)
  Week 4: Head/Neck Scaling (n=47, 47, 48, 46) | 1.5 (0.16) | 1.1 (0.15) | 0.9 (0.14) | 1.8 (0.16)
  Week 4: Upper Limbs Scaling (n=47, 47, 48, 46) | 2.0 (0.12) | 1.9 (0.16) | 1.6 (0.14) | 2.3 (0.11)
  Week 4: Trunk Scaling (n=47, 47, 48, 46) | 1.8 (0.15) | 1.5 (0.16) | 1.4 (0.12) | 2.4 (0.12)
  Week 4: Lower Limbs Scaling (n=47, 47, 48, 46) | 2.4 (0.11) | 2.0 (0.15) | 1.8 (0.14) | 2.5 (0.12)
  Week 8: Head/Neck Scaling (n=43, 40, 47, 39) | 1.2 (0.15) | 0.8 (0.16) | 0.7 (0.14) | 1.6 (0.16)
  Week 8: Upper Limbs Scaling (n=43, 40, 47, 39) | 1.7 (0.14) | 1.5 (0.16) | 1.3 (0.14) | 2.2 (0.15)
  Week 8: Trunk Scaling (n=43, 40, 47, 39) | 1.4 (0.16) | 1.2 (0.19) | 1.0 (0.14) | 2.1 (0.13)
  Week 8: Lower Limbs Scaling (n=43, 40, 47, 39) | 1.9 (0.16) | 1.5 (0.16) | 1.3 (0.15) | 2.4 (0.15)
  Week 12: Head/Neck Scaling (n=38, 39, 43, 34) | 1.0 (0.17) | 0.8 (0.14) | 0.5 (0.12) | 1.6 (0.18)
  Week 12: Upper Limbs Scaling (n=38, 39, 43, 34) | 1.5 (0.16) | 1.4 (0.13) | 1.1 (0.14) | 2.0 (0.18)
  Week 12: Trunk Scaling (n=38, 39, 43, 34) | 1.3 (0.18) | 1.0 (0.18) | 0.7 (0.12) | 1.9 (0.19)
  Week 12: Lower Limbs Scaling (n=38, 39, 43, 34) | 1.8 (0.18) | 1.4 (0.14) | 0.9 (0.13) | 2.3 (0.18)
  Week 14: Head/Neck Scaling (n=38, 37, 37, 33) | 1.2 (0.18) | 1.1 (0.19) | 0.9 (0.18) | 1.7 (0.18)
  Week 14: Upper Limbs Scaling (n=38, 37, 37, 33) | 1.8 (0.16) | 1.6 (0.15) | 1.3 (0.17) | 2.1 (0.17)
  Week 14: Trunk Scaling (n=38, 37, 37, 33) | 1.5 (0.18) | 1.3 (0.18) | 1.1 (0.18) | 1.8 (0.18)
  Week 14: Lower Limbs Scaling (n=38, 37, 37, 33) | 1.9 (0.18) | 1.5 (0.16) | 1.3 (0.20) | 2.2 (0.19)
  Week 16: Head/Neck Scaling (n=37, 36, 41, 30) | 1.2 (0.19) | 1.6 (0.20) | 1.0 (0.17) | 1.7 (0.22)
  Week 16: Upper Limbs Scaling (n=37, 36, 41, 30) | 1.9 (0.19) | 1.7 (0.16) | 1.7 (0.16) | 2.3 (0.18)
  Week 16: Trunk Scaling (n=37, 36, 41, 30) | 1.7 (0.20) | 1.5 (0.18) | 1.4 (0.16) | 2.0 (0.20)
  Week 16: Lower Limbs Scaling (n=37, 36, 41, 30) | 2.2 (0.19) | 1.8 (0.17) | 1.5 (0.17) | 2.4 (0.19)
  Baseline: PASI Total Score | 21.5 (0.97) | 21.2 (1.15) | 22.6 (1.49) | 21.5 (1.01)
  Week 2: PASI Total Score | 17.0 (0.97) | 16.3 (1.39) | 15.3 (1.27) | 20.4 (1.23)
  Week 4: PASI Total Score | 14.0 (0.98) | 12.3 (1.46) | 10.4 (1.13) | 19.1 (1.50)
  Week 8: PASI Total Score | 10.7 (1.02) | 8.1 (1.45) | 6.9 (1.14) | 17.3 (1.31)
  Week 12: PASI Total Score | 9.6 (1.18) | 5.7 (0.73) | 5.0 (0.87) | 15.8 (1.30)
  Week 14: PASI Total Score | 10.8 (1.18) | 7.6 (1.06) | 6.7 (1.37) | 16.1 (1.39)
  Week 16: PASI Total Score | 11.9 (1.33) | 9.1 (0.91) | 8.8 (1.26) | 16.4 (1.66)

7. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Component Scores and Total Score at Week 2, 4, 8, 12, 14, and 16
Description: as for outcome 1
Time Frame: Baseline, Week 2, 4, 8, 12, 14, 16
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 48 | 50
units on a scale
  Week 2: Head/Neck Erythema (n=47, 48, 48, 49) | -0.4 (0.10) | -0.7 (0.13) | -1.0 (0.15) | -0.2 (0.08)
  Week 2: Upper Limbs Erythema (n=47, 48, 48, 49) | -0.6 (0.11) | -0.5 (0.09) | -0.8 (0.10) | -0.2 (0.09)
  Week 2: Trunk Erythema (n=47, 48, 48, 49) | -0.6 (0.12) | -0.6 (0.12) | -0.8 (0.13) | -0.2 (0.10)
  Week 2: Lower Limbs Erythema (n=47, 48, 48, 49) | -0.4 (0.11) | -0.6 (0.11) | -0.8 (0.11) | -0.2 (0.09)
  Week 4: Head/Neck Erythema (n=47, 47, 48, 46) | -0.7 (0.13) | -1.0 (0.15) | -1.4 (0.16) | -0.3 (0.15)
  Week 4: Upper Limbs Erythema (n=47, 47, 48, 46) | -0.9 (0.14) | -1.0 (0.11) | -1.3 (0.12) | -0.5 (0.09)
  Week 4: Trunk Erythema (n=47, 47, 48, 46) | -0.9 (0.14) | -0.8 (0.12) | -1.3 (0.12) | -0.4 (0.07)
  Week 4: Lower Limbs Erythema (n=47, 47, 48, 46) | -0.7 (0.13) | -0.9 (0.11) | -1.3 (0.12) | -0.4 (0.09)
  Week 8: Head/Neck Erythema (n=43, 40, 47, 39) | -1.0 (0.14) | -1.3 (0.19) | -1.7 (0.18) | -0.6 (0.18)
  Week 8: Upper Limbs Erythema (n=43, 40, 47, 39) | -1.2 (0.16) | -1.2 (0.14) | -1.7 (0.14) | -0.6 (0.10)
  Week 8: Trunk Erythema (n=43, 40, 47, 39) | -1.1 (0.18) | -1.2 (0.15) | -1.7 (0.17) | -0.5 (0.12)
  Week 8: Lower Limbs Erythema (n=43, 40, 47, 39) | -1.1 (0.16) | -1.4 (0.16) | -1.8 (0.16) | -0.5 (0.10)
  Week 12: Head/Neck Erythema (n=38, 39, 43, 34) | -1.1 (0.17) | -1.2 (0.18) | -2.0 (0.19) | -0.6 (0.20)
  Week 12: Upper Limbs Erythema (n=38, 39, 43, 34) | -1.3 (0.17) | -1.3 (0.14) | -1.8 (0.15) | -0.7 (0.14)
  Week 12: Trunk Erythema (n=38, 39, 43, 34) | -1.2 (0.20) | -1.3 (0.19) | -1.9 (0.18) | -0.5 (0.18)
  Week 12: Lower Limbs Erythema (n=38, 39, 43, 34) | -1.2 (0.18) | -1.5 (0.14) | -1.9 (0.17) | -0.4 (0.12)
  Week 14: Head/Neck Erythema (n=38, 37, 37, 33) | -1.0 (0.18) | -1.0 (0.19) | -1.5 (0.21) | -0.6 (0.19)
  Week 14: Upper Limbs Erythema (n=38, 37, 37, 33) | -1.1 (0.17) | -1.0 (0.17) | -1.5 (0.18) | -0.7 (0.13)
  Week 14: Trunk Erythema (n=38, 37, 37, 33) | -1.1 (0.19) | -1.0 (0.20) | -1.6 (0.20) | -0.5 (0.18)
  Week 14: Lower Limbs Erythema (n=38, 37, 37, 33) | -1.1 (0.16) | -1.2 (0.17) | -1.6 (0.20) | -0.4 (0.14)
  Week 16: Head/Neck Erythema (n=37, 36, 41, 30) | -0.9 (0.19) | -0.5 (0.18) | -1.3 (0.21) | -0.5 (0.22)
  Week 16: Upper Limbs Erythema (n=37, 36, 41, 30) | -0.8 (0.19) | -0.7 (0.16) | -1.0 (0.17) | -0.6 (0.14)
  Week 16: Trunk Erythema (n=37, 36, 41, 30) | -0.9 (0.22) | -0.6 (0.17) | -1.1 (0.20) | -0.6 (0.19)
  Week 16: Lower Limbs Erythema (n=37, 36, 41, 30) | -0.7 (0.18) | -1.0 (0.18) | -1.3 (0.18) | -0.4 (0.13)
  Week 2: Head/Neck Induration (n=47, 48, 48, 49) | -0.6 (0.11) | -0.4 (0.11) | -0.8 (0.13) | -0.2 (0.09)
  Week 2: Upper Limbs Induration (n=47, 48, 48, 49) | -0.5 (0.09) | -0.5 (0.08) | -0.8 (0.11) | -0.1 (0.09)
  Week 2: Trunk Induration (n=47, 48, 48, 49) | -0.4 (0.10) | -0.6 (0.11) | -0.6 (0.11) | -0.3 (0.07)
  Week 2: Lower Limbs Induration (n=47, 48, 48, 49) | -0.3 (0.08) | -0.4 (0.08) | -0.7 (0.12) | -0.2 (0.09)
  Week 4: Head/Neck Induration (n=47, 47, 48, 46) | -0.8 (0.11) | -0.9 (0.13) | -1.3 (0.16) | -0.3 (0.15)
  Week 4: Upper Limbs Induration (n=47, 47, 48, 46) | -0.6 (0.12) | -0.8 (0.12) | -1.3 (0.13) | -0.3 (0.10)
  Week 4: Trunk Induration (n=47, 47, 48, 46) | -0.8 (0.12) | -0.7 (0.13) | -1.2 (0.12) | -0.4 (0.10)
  Week 4: Lower Limbs Induration (n=47, 47, 48, 46) | -0.6 (0.12) | -0.8 (0.12) | -1.2 (0.13) | -0.5 (0.10)
  Week 8: Head/Neck Induration (n=43, 40, 47, 39) | -1.0 (0.13) | -1.1 (0.16) | -1.5 (0.18) | -0.5 (0.14)
  Week 8: Upper Limbs Induration (n=43, 40, 47, 39) | -0.9 (0.15) | -1.1 (0.13) | -1.5 (0.16) | -0.3 (0.12)
  Week 8: Trunk Induration (n=43, 40, 47, 39) | -1.0 (0.16) | -1.1 (0.16) | -1.5 (0.15) | -0.6 (0.13)
  Week 8: Lower Limbs Induration (n=43, 40, 47, 39) | -1.0 (0.15) | -1.3 (0.16) | -1.6 (0.17) | -0.5 (0.10)
  Week 12: Head/Neck Induration (n=38, 39, 43, 34) | -1.2 (0.16) | -1.2 (0.15) | -1.7 (0.18) | -0.4 (0.17)
  Week 12: Upper Limbs Induration (n=38, 39, 43, 34) | -1.2 (0.15) | -1.2 (0.13) | -1.6 (0.17) | -0.5 (0.16)
  Week 12: Trunk Induration (n=38, 39, 43, 34) | -1.1 (0.18) | -1.2 (0.14) | -1.8 (0.16) | -0.7 (0.15)
  Week 12: Lower Limbs Induration (n=38, 39, 43, 34) | -1.2 (0.16) | -1.4 (0.15) | -1.7 (0.15) | -0.5 (0.11)
  Week 14: Head/Neck Induration (n=38, 37, 37, 33) | -1.1 (0.15) | -0.8 (0.16) | -1.4 (0.20) | -0.5 (0.17)
  Week 14: Upper Limbs Induration (n=38, 37, 37, 33) | -0.8 (0.15) | -1.0 (0.16) | -1.4 (0.18) | -0.5 (0.16)
  Week 14: Trunk Induration (n=38, 37, 37, 33) | -1.0 (0.18) | -0.9 (0.15) | -1.5 (0.20) | -0.7 (0.17)
  Week 14: Lower Limbs Induration (n=38, 37, 37, 33) | -1.1 (0.16) | -1.1 (0.18) | -1.4 (0.20) | -0.5 (0.13)
  Week 16: Head/Neck Induration (n=37, 36, 41, 30) | -1.1 (0.15) | -0.4 (0.18) | -1.3 (0.20) | -0.3 (0.19)
  Week 16: Upper Limbs Induration (n=37, 36, 41, 30) | -0.8 (0.17) | -0.6 (0.16) | -1.2 (0.18) | -0.4 (0.18)
  Week 16: Trunk Induration (n=37, 36, 41, 30) | -0.9 (0.20) | -0.6 (0.14) | -1.1 (0.19) | -0.6 (0.18)
  Week 16: Lower Limbs Induration (n=37, 36, 41, 30) | -1.0 (0.19) | -0.8 (0.16) | -1.4 (0.18) | -0.4 (0.14)
  Week 2: Head/Neck Scaling (n=47, 48, 48, 49) | -0.5 (0.12) | -0.6 (0.13) | -0.9 (0.13) | -0.3 (0.09)
  Week 2: Upper Limbs Scaling (n=47, 48, 48, 49) | -0.4 (0.10) | -0.6 (0.10) | -0.6 (0.10) | -0.2 (0.08)
  Week 2: Trunk Scaling (n=47, 48, 48, 49) | -0.3 (0.12) | -0.6 (0.13) | -0.7 (0.11) | -0.2 (0.10)
  Week 2: Lower Limbs Scaling (n=47, 48, 48, 49) | -0.4 (0.10) | -0.4 (0.09) | -0.6 (0.11) | -0.2 (0.09)
  Week 4: Head/Neck Scaling (n=47, 47, 48, 46) | -0.7 (0.14) | -1.0 (0.15) | -1.4 (0.15) | -0.4 (0.14)
  Week 4: Upper Limbs Scaling (n=47, 47, 48, 46) | -0.5 (0.14) | -0.8 (0.12) | -1.0 (0.13) | -0.3 (0.10)
  Week 4: Trunk Scaling (n=47, 47, 48, 46) | -0.6 (0.13) | -0.9 (0.13) | -1.1 (0.14) | -0.2 (0.09)
  Week 4: Lower Limbs Scaling (n=47, 47, 48, 46) | -0.7 (0.09) | -0.9 (0.12) | -0.9 (0.14) | -0.4 (0.11)
  Week 8: Head/Neck Scaling (n=43, 40, 47, 39) | -1.0 (0.19) | -1.4 (0.19) | -1.6 (0.18) | -0.4 (0.16)
  Week 8: Upper Limbs Scaling (n=43, 40, 47, 39) | -0.8 (0.16) | -1.2 (0.13) | -1.3 (0.16) | -0.4 (0.14)
  Week 8: Trunk Scaling (n=43, 40, 47, 39) | -1.0 (0.18) | -1.2 (0.16) | -1.5 (0.17) | -0.5 (0.12)
  Week 8: Lower Limbs Scaling (n=43, 40, 47, 39) | -1.1 (0.14) | -1.3 (0.15) | -1.4 (0.15) | -0.5 (0.13)
  Week 12: Head/Neck Scaling (n=38, 39, 43, 34) | -1.2 (0.19) | -1.4 (0.19) | -1.8 (0.18) | -0.3 (0.20)
  Week 12: Upper Limbs Scaling (n=38, 39, 43, 34) | -1.0 (0.18) | -1.3 (0.14) | -1.5 (0.17) | -0.6 (0.17)
  Week 12: Trunk Scaling (n=38, 39, 43, 34) | -1.2 (0.19) | -1.4 (0.17) | -1.8 (0.16) | -0.7 (0.17)
  Week 12: Lower Limbs Scaling (n=38, 39, 43, 34) | -1.3 (0.15) | -1.4 (0.15) | -1.7 (0.15) | -0.6 (0.15)
  Week 14: Head/Neck Scaling (n=38, 37, 37, 33) | -1.0 (0.19) | -1.0 (0.19) | -1.4 (0.20) | -0.3 (0.18)
  Week 14: Upper Limbs Scaling (n=38, 37, 37, 33) | -0.7 (0.16) | -1.1 (0.17) | -1.3 (0.18) | -0.6 (0.16)
  Week 14: Trunk Scaling (n=38, 37, 37, 33) | -0.8 (0.18) | -1.0 (0.16) | -1.4 (0.20) | -0.8 (0.17)
  Week 14: Lower Limbs Scaling (n=38, 37, 37, 33) | -1.2 (0.17) | -1.2 (0.17) | -1.4 (0.19) | -0.7 (0.16)
  Week 16: Head/Neck Scaling (n=37, 36, 41, 30) | -1.0 (0.18) | -0.5 (0.18) | -1.4 (0.20) | -0.2 (0.22)
  Week 16: Upper Limbs Scaling (n=37, 36, 41, 30) | -0.7 (0.16) | -1.0 (0.14) | -1.0 (0.16) | -0.5 (0.18)
  Week 16: Trunk Scaling (n=37, 36, 41, 30) | -0.8 (0.20) | -0.8 (0.15) | -1.2 (0.19) | -0.7 (0.19)
  Week 16: Lower Limbs Scaling (n=37, 36, 41, 30) | -0.9 (0.16) | -0.9 (0.18) | -1.2 (0.19) | -0.6 (0.17)
  Week 2: PASI Total Score (n=47, 48, 48, 49) | -4.7 (0.81) | -4.7 (0.62) | -7.3 (0.86) | -0.8 (0.69)
  Week 4: PASI Total Score (n=47, 47, 48, 46) | -7.5 (1.05) | -8.6 (0.93) | -12.2 (1.18) | -2.7 (0.86)
  Week 8: PASI Total Score (n=43, 40, 47, 39) | -10.9 (1.41) | -11.6 (1.09) | -15.8 (1.38) | -3.7 (0.96)
  Week 12: PASI Total Score (n=38, 39, 43, 34) | -12.1 (1.59) | -13.1 (1.05) | -17.9 (1.59) | -5.1 (1.16)
  Week 14: PASI Total Score (n=38, 37, 37, 33) | -10.9 (1.58) | -11.4 (1.13) | -16.5 (1.95) | -4.4 (1.32)
  Week 16: PASI Total Score (n=37, 36, 41, 30) | -9.7 (1.57) | -9.3 (1.09) | -14.0 (1.77) | -5.1 (1.42)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 2 mg | CP-690,550 5 mg | CP-690,550 15 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/49 | 1/49 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 25/49 | 28/49 | 30/49 | 30/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 2 mg (N=49) | CP-690,550 5 mg (N=49) | CP-690,550 15 mg (N=49) | Placebo (N=50)
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 2 mg (N=49) | CP-690,550 5 mg (N=49) | CP-690,550 15 mg (N=49) | Placebo (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2
Hernia (General disorders) | 0 | 1 | 0 | 0
Therapeutic response unexpected (General disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 2
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3 | 5
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 5 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 2 | 5
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0
Cytomegalovirus test positive (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 1 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 4 | 3 | 3 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 4
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Endodontic procedure (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.